CLINICAL TRIAL: NCT07054554
Title: Engaging Mental Health Services for Preschoolers at Risk
Acronym: NTRI-MH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelly Kamimura-Nishimura, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R34MH137224-01 (NIH); R34MH137224 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-07-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Disorder; Family Navigation; Minoritized Population; Preschool Age Children
Keywords: Family Navigation; mental health disorder; Preschool Age Children
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: NTRI-MH intervention will use evidence-based instructional strategies for adult professional development (i.e., lecture, discussion, case studies, role-playing). NTRI-MH training includes 20 hours of didactic and interactive sessions (5 sessions of 4 hours each) covering the following areas specific to MH needs in young children at-risk: 1) benefits and barriers (professional and family) to early intervention for children with MH concerns, 2) approaches for empowering caregivers, 3) supporting strategies to assist families through early MH access and service engagement, 4) use of the dashboard to track and monitor the course of clinical, functional, and behavioral outcomes, 5) evidence-based working alliances with PCPs and teachers (including a 2-hour session with the child's teacher), and 6) MH resources, treatments and services, and strategies to support parental management of young child behaviors.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (NTRI-MH) (Experimental): For the intervention group, the navigators will implement the NTRI-MH for 6 months with the caregivers, including 15 hours of navigation services with a 2-hour face-to-face meeting, at least 3 monthly in-person meetings, attending assessments and treatments with the caregivers at HStart, PCP offices, and MH services locations. After these visits, the navigator will follow up by phone, text, or email with the caregiver. Navigators will meet weekly with research staff for supervision and case review. Teachers will share a copy of screenings and recommend a visit with PCP, and PCPs will review the Just-In-Time packet and make referrals.
  Interventions: Other: NTRI-MH
- Control (No Intervention): The caregivers in the active control group will receive a 2-hour training seminar and educational materials including handouts/videos from a developmental activities' toolkit pertinent to the emotional, behavioral, and developmental age of their child. The training seminar will include topics of common MH concerns of young children, steps to addressing challenging behavior, strategies for decreasing problems behaviors, and crisis management.

INTERVENTIONS:
Other: NTRI-MH — NTRI-MH intervention will use evidence-based instructional strategies for adult professional development (i.e., lecture, discussion, case studies, role-playing). NTRI-MH training includes 20 hours of didactic and interactive sessions (5 sessions of 4 hours each) covering the following areas specific to MH needs in young children at-risk: 1) benefits and barriers (professional and family) to early intervention for children with MH concerns, 2) approaches for empowering caregivers, 3) supporting strategies to assist families through early MH access and service engagement , 4) use of the dashboard to track and monitor the course of clinical, functional, and behavioral outcomes, 5) evidence-based working alliances with PCPs and teachers (including a 2 hour session with the child's teacher), and 6) MH resources, treatments and services, and strategies to support parental management of young child behaviors.
  Arms: Intervention (NTRI-MH)

SUMMARY:
Most mental health (MH) disorders develop in early childhood but are not clinically identified or treated until later-delaying treatment services that could prevent the enduring effects of long-term MH problems. Moreover, low income, ethno-racial minoritized children who exhibit higher rates of persistent MH disorders, are at greater risk for lags in identification and treatment. Head Start (HStart) has shown early school success for low-income children, aged 3-5 years, who are disproportionately Black or Latinx. HStart monitors early childhood MH symptoms, yet studies have found that when detected, only those most impaired are referred for treatment. In our research, the investigators learned that system and individual level barriers preclude early treatment among HStart preschoolers with developmental concern. The investigators showed that caregivers encountered system barriers of HStart teachers and primary care providers (PCPs) falling behind in referrals for intervention, and caregiver beliefs about stigma, their limited knowledge and distrust of healthcare hindered early engagement in services. Studies on MH treatment obstacles for low-income, ethno-racial minoritized people illustrate similar barriers to those found among HStart preschoolers with developmental concern. We developed and tested an ethno-racially matched, peer-based family navigator program for HStart preschoolers with developmental concern. Navigators used trust and empowerment to increase caregiver advocacy thereby leading to improved professional alliances and treatment. A navigator program for those with primary MH concerns has not been trialed. For Aim 1, the investigators aim to tailor and trial in a case series the Navigate-Train-Referral-Intervention Mental Health (NTRI-MH) intervention to promote access, engagement, coordination, and optimization of services for preschoolers with MH symptoms. The investigators have used focus group feedback from caregiver, navigator, HStart teacher, and PCP stakeholders to adapt NTRI-MH and created a web-based dashboard to monitor outcomes (Phase 1). Then, for phase 2, the investigators will conduct a feasibility study for caregivers of HStart preschoolers with MH symptoms, guided by ethno-racially matched family navigators and referrals by HStart teachers and PCPs (n=20). Further, for Aim 2, the investigators will pilot test NTRI-MH for caregivers of preschoolers with MH symptoms compared to an active control group of caregivers who receive child behavior training (n=86). The investigators will trial the effectiveness of the NTRI-MH mechanisms of caregiver beliefs on MH, empowerment, and professional alliances on family functioning and child emotion regulation. If the aims of the project are achieved, this study would have a large impact on early MH service use for ethno-racial minoritized young children with the potential to improve child MH outcomes.

DETAILED DESCRIPTION:
The proposed project involves three phases:

Aim 1 (Phase 1): Focus groups. Six focus groups will be held to elucidate barriers and facilitators to access and engagement of HStart children in MH services. Separate focus groups will be conducted for each stakeholder and ethno-racial caregiver group (3 Black, Latinx, and White caregiver groups, 1 navigator, 1 teacher, and 1 PCP focus group). Latinx caregivers and navigators will have the option to attend an English or Spanish focus group session. The focus groups will be conducted via a web-based platform (e.g., MS Teams) at a variety of times to facilitate participation of caregivers, navigators, and professionals who provide childcare and/or work at different times or lack transportation or childcare to attend in-person sessions. Demographic data will be collected. Groups will employ an open format with guided questions to gain perspective and to help participants focus on 1) barriers and facilitators to access and engagement in MH services, 2) enriching a navigation program to address MH barriers and enhance facilitators, and 3) conceptualize the ideal dashboard to track and monitor the trajectory of MH clinical, functional, and behavioral outcomes. To ensure research integrity, focus group facilitation will be led by the co-PIs and research team experienced with focus groups. All sessions will be recorded, field notes composed, and sessions transcribed verbatim.

Web-based dashboard. The investigators will develop a web-based dashboard on a secure website to assist the navigators, and us, the research team, in monitoring and tracking child and caregiver progress over time with clinical, functional, and behavioral outcomes. This user-friendly system will track and monitor alignment of caregiver goals to service use on the primary outcomes of access, engagement, coordination, and optimization of MH services. Also, it will track the child's MH symptoms in the case series and pilot study. The goals and tasks will be set by the caregiver and navigator after visits with professionals, maximizing the benefits of goal-setting that include motivation, commitment, and self-regulation and working professional alliances. The research team will rate the progress toward the caregiver-determined goals and the child's MH symptoms from the data will allow us to measure care coordination. Access data on detection of risk for MH disorder and appropriateness of referrals will be inputted from the HStart data base (ChildPlus©), medical record, and navigator tracking of visits and referrals by teachers and PCPs and recommendations made. Engagement will be monitored by caregiver/navigator meeting content and goals, caregiver goal alignment with professional recommendations, and resources/tasks needed to reach the goals. Coordination will be tracked with caregiver initiation, completion and frequency of the child's MH services, and navigator-provided resources on advocacy, emotional support, basic needs, and MH disorders to support services use. Optimization will be monitored by agreement between caregivers and PCPs on the MH treatment goals and tasks including services type and frequency. The dashboard will be a core component of the NTRI-MH treatment manual. It will be built with the capacity to eventually scale up to involve caregivers, teachers, and PCPs in monitoring and tracking the trajectory of progress over time.

NTRI-MH adaptation. The stakeholder focus group findings and views on dashboard creation will inform the modifications to the 1st iteration of the NTRI-MH treatment manual. Adaptations to the treatment manual will focus on the barriers and facilitators to engagement in MH services, navigation enhancements to address these barriers, usefulness of the dashboard to track and monitor progress in MH outcomes. Implementation fidelity questionnaires will be modified for NTRI-MH. Once the NTRI-MH treatment manual is revised, the full research team and consultants will review it for a 2nd iteration. The NTRI-MH treatment manual adaptations will be completed prior to being implemented in the case series trial.

The primary deliverable is modification of the NTRI-MH intervention design and the content of a web-based dashboard to adapt the treatment manual for addressing the primary outcomes of access, engagement, coordination, and optimization of MH services.

Aim 1 (Phase 2): NTRI-MH training and implementation. Training for the navigators and teachers will use evidence-based instructional strategies for adult professional development (i.e., lecture, discussion, case studies, role-playing).92 PCPs will receive training when their patient enters the study. The research team will provide training for the navigators and teachers, whereas the PCPs will receive training by e-Learning. Since the navigators were previously trained in NTRI-DD, navigators training will be adjusted to include adaptations to the NTRI-MH implementation and treatment manual, and use of the dashboard to assist navigation. This comprises 20 hours of didactic and interactive sessions (5 sessions of 4 hours each). The navigators' NTRI-MH training will include these areas specific to MH needs in young children at-risk: 1) benefits and barriers (professional and family) to early intervention for children with MH concerns, 2) approaches for empowering caregivers, 3) supporting strategies to assist families through early MH access and service engagement , 4) use of the dashboard to track and monitor the course of clinical, functional, and behavioral outcomes, 5) evidence-based working alliances with PCPs and teachers (including a 2 hour session with the child's teacher), and 6) MH resources, treatments and services, and strategies to support parental management of young child behaviors (See Appendix A). Teacher training will encompass 5 hours of didactic and interactive sessions with continuing education credits and focus on: 1) delivering difficult news to families of children at-risk for MH and use of letter for explaining screenings and next steps, 2) strategies to recommend the child visit their PCP for MH concerns, 3) evidence-based working alliances with caregivers, PCPs, and navigators (including a 2-hour session with the caregiver's navigators). PCP training will be formatted as 1-hour e-Learning with continuing education credit and focus on: 1) acting early to manage and mitigate MH disorders and use of the Just-In-Time decision aid, 2) talking to caregivers about evidence-based and appropriate treatments and services for MH, and 4) evidence-based working alliances with caregivers, teachers, and navigators. All training will be evaluated at the final training sessions. Following training, NTRI-MH implementation will comprise navigators executing the 3-month NTRI-MH intervention with the caregivers, including 10 hours of navigation services with a 1-to-2-hour face-to-face meeting, at least 3 monthly in-person meetings, and attending all meetings, visits, and/or services with the caregivers at HStart, primary care offices, and MH centers. After each visit, the navigator will follow up by phone, text, or e-mail with the caregiver and review goals and tasks and enter the dashboard data. Navigators will meet weekly with research staff for supervision and case review. Teachers will share a copy of the screenings with caregivers, a letter explaining the screening results, and recommend a visit with the child's PCP. PCPs will complete the e-Learning session, review the Just-In-Time decision aid (i.e., child's screening results and evidence-based treatment recommendations), and make referrals. Navigators, caregivers, teachers, and PCPs will complete questionnaires at baseline (Time 1), immediately post-intervention (Time 2), and 3-months post-intervention (Time 3). The study team will assess the child's MH symptoms and family function at baseline, post-intervention, and 3-months following. Findings from the assessments obtained at times 1, 2, and 3 will inform ongoing modifications to the NTRI-MH dashboard and treatment manual, and the dashboard evaluated by the navigators at a final weekly supervision meeting. In addition, at the end of the case series feasibility study the co-PIs will interview the navigators and caregivers to gain a more detailed understanding of their NTRI-MH experiences and the descriptive data compiled for treatment manual revisions.

Aim 1 (Phase 2) study measures include primary outcomes (NTRI-MH's feasibility and implementation by navigators; NTRI-MH satisfaction as per caregivers, navigators, teachers, and PCPs) and potential mechanisms of action (beliefs/perceptions about MH and its treatment, feelings of empowerment, working alliance with professionals) effects on access, engagement, coordination, and optimization of MH services and the child's MH symptoms and family function. The primary deliverable is a modified dashboard and NTRI-MH treatment manual with high feasibility, acceptability, and implementation ratings, and a preliminary description of a trend showing the potential mechanisms of action affect access, engagement, coordination, and optimization of MH services for at-risk preschoolers and the downstream outcomes of family function and the child's MH symptoms.

Aim 2: Ten navigators will implement the NTRI-MH. Caregivers will be randomly assigned by schools to the intervention group (n=30) or control group (n=30). Navigators', teachers', and PCPs' training will follow procedures outlined in Aim 1 (Phase 2), except for 10 additional training hours for all navigators to allow for changes needed since the treatment manual revisions. Following training, for the intervention group, the navigators will implement the NTRI-MH for 6 months with the caregivers, including 15 hours of navigation services with a 2-hour face-to-face meeting, at least 6 monthly in-person meetings, attending assessments and treatments with the caregivers at HStart, PCP offices, and MH services locations. After these visits, the navigator will follow up by phone, text, or email with the caregiver. Navigators will meet weekly with research staff for supervision and case review. Teachers will share a copy of screenings and recommend a visit with PCP, and PCPs will review the Just-In-Time packet and make referrals. The caregivers in the active control group will receive a 2-hour training seminar and educational materials including handouts and videos from a developmental activities' toolkit pertinent to the emotional, behavioral, and developmental age of their child. Navigators, caregivers, teachers, and PCPs from both the intervention and control groups will complete questionnaires at baseline (Time 1), immediately post-intervention (Time 2), and 3 months post-intervention (Time 3). The NTRI-MH treatment manual will be modified from analysis of the assessments and expert feedback solicited to create the final NTRI-MH treatment manual and R01 application revised accordingly.

NTRI-MH measures will be identical for both the intervention and control groups, except for intervention feasibility, acceptability, and implementation. Table 3 describes Aim 2 study measures, including primary outcomes (access, engagement, coordination, and optimization of MH services) and secondary outcomes (child's MH symptoms, family functioning, NTRI-MH acceptability, feasibility, and implementation). We will also measure potential mechanisms of action (beliefs/perceptions about MH and its treatment, feelings of empowerment, working alliance with professionals) to determine if these improve access, engagement, coordination, and optimization of MH services for at-risk preschoolers. The primary deliverable is revisions to NRTI-MH and dashboard in a treatment manual that attends to potential mechanisms impacting access, engagement, coordination, and optimization of MH services in at-risk preschoolers, child/caregiver outcomes and preliminary data to inform larger efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

* Family Navigators: Having experience working as family navigator and/or community health worker; Latinx, Black or White; > 18 years old.
* Caregivers: current caregiver of a HStart preschooler at-risk for MH disorders (ASQ-SE above threshold score)
* Teachers: Current Head Start (HStart) teacher from one of the 2 HStart site;> 18 years old; Any race/ethnicity.
* PCPs: Currently providing primary care for HStart preschool age children at risk for MH disorders; > 18 years old; Any race/ethnicity.

Exclusion Criteria:

* Unable to read/speak either English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Navigate-Train-Referral-Intervention-Mental-Health (NTRI-MH) Satisfaction Questionnaire | Immediately after intervention and 3 months after intervention
  This is a 7-item Likert scale questionnaire that elicits caregivers' and family navigators' opinions regarding the format, content, length, and convenience of the intervention.
  Score Range: 7-28 (the higher the score, better satisfaction)
System Usability Scale | Immediately after intervention and 3-months after intervention
  The SUS is a 10-item Likert scale questionnaire that elicits family navigators', teachers', and PCPs' global views of the NTRI-MH treatment manual's usability.
  Score range: 0-100 (the higher the score, better usability)
Family Navigator Activities Checklist | 3-months after intervention
  This 29-item checklist will document family navigator-caregiver activities, including emotional support, action planning, information provision, advocacy, and skill development.
  Range 0-29 (the higher the score, more activities completed)
Implementation Questionnaire | 3-months after intervention
  The implementation questionnaire will include 12-Likert score items recording information about acceptability, intervention appropriateness and feasibility of the intervention.
  Score range: 12-60 (the higher the score, better acceptability, feasibility, and appropriateness)
Referrals to Primary Care Providers (PCPs) and mental health services | Baseline
  We will obtain data regarding referrals made to PCPs and/or mental health services by Head Start teachers though reviewing the ChildPlus Head Start Database.
Referrals to mental health services | Immediately after intervention and 3-months after intervention
  We will obtain data regarding referrals to mental health services by Primary Care Providers (PCPs) through medical chart review.
Access to mental health services | Baseline, immediately after intervention, and 3-months after intervention
  Using a web-based electronic dashboard, user-friendly system, we will record the number of referrals to mental health services.
Parental Stress Scale | Baseline, immediately after intervention, and 3-months after intervention
  This is an 18-item self-report measure in which parents respond to statements about their typical relationship with their child. This measure will assess parents' feelings about positive aspects (e.g., emotional benefits, personal development) and negative views of parenting (e.g., demands on resources, feelings of stress). The possible range of PSS is 18 (low stress) to 90 (high stress).
Engagement and coordination to mental health services | Baseline, after intervention, 3-months after intervention
  Using a web-based electronic dashboard, we will record the alignment with mental health recommendations.
Optimization of mental health services | Baseline, immediately after intervention, 3-months after intervention
  Using a web-based, electronic dashboard, we will record the caregiver agreement with goals and tasks.

OTHER OUTCOMES:
Brief Illness Perceptions Questionnaire | Baseline, immediately after intervention, and 3-months after intervention
  This 11-item scale is designed to assess a parent's representation of mental health disorders (e.g. expected time course, consequences, causes, etc.). It has good test-retest reliability as well as concurrent and predictive validity. All of the items, except the causal scale, are rated using a 0 to 10 response scale. For the causal scale, parents list the three most important causal factors in their child's mental health disorder, and responses are grouped into categories (genetic, environmental, behavioral, dietary, etc.) for analysis.
Decisional Conflict Scale | Baseline, immediately after intervention, and 3-months after intervention
  This 16-item validated measure elicits the parent's preference for treatment options and parent perceived sources of decisional conflict about their preferred option. The scale produces a total score with five subscales: 1) informed; 2) values clarity; 3) support; 4) uncertainty; 5) effective decision. Lower scores are desirable, with a range from 0-100.
Family Empowerment Scale | Baseline, immediately after intervention, 3-months after intervention
  The FES is a 12-item scale that assess perceptions and attitudes about family navigator and caregiver roles/responsibilities within their local service systems and their ability to advocate on behalf of their children. Items are scored on a 5-point likert type scale from 1 (Never) to 5 (Very often). The FES assesses three domains, Work (e.g. "I know what to do when problems arise with the families with whom I work"), Children's Services (e.g., "I make sure that professionals understand caregivers' opinions about what services their children need"), and Community (e.g. "I feel I can have a part in improving services for children in my community")
Collaborative Skills Questionnaire | Baseline, immediately after intervention, 3-months after intervention
  The CSQ is a 36-item scale examining key knowledge and skills development related to training modules. It includes six subscales, one for each I2-ART training manual module: (1) Listening, Engagement, and Boundary Settings Skills, (2) Group Management, (3) Priority Setting, (4) Specific Disorders and Their Treatment, (5) Mental Health Services, and (6) School Options. Questions include, "I can talk to parents about our mutual responsibilities in the working relationship" and "I am aware of barriers that parents may face in seeking help for their children and know how to help them overcome those barriers."
Vanderbilt Mental Health Services Efficacy | Baseline, immediately after intervention, and 3 months after intervention
  This 25-item scale examines the degree to which family navigators and caregivers feel effective in accessing mental health services. Items are scored on a five-point scale from 1 (strongly disagree) to 5 (strongly agree). Typical items include, "I believe that I can help parents access and use effectively mental health services for their children" and "My skills in dealing with mental health services will help me to empower parents to change things that might be wrong with their child's treatment."
Working Alliance Inventory | Baseline, immediately after intervention, and 3 months after intervention
  The WAI is a 12-item measure of a family's perceived agreement with their healthcare provider on the goals/tasks of treatment and the extent to which they have a strong personal bond with their provider. Respondents rate their responses on a scale of 1 (strongly disagree) to 5 (strongly agree). Item scores are summed, giving a range from 12-60, with higher scores indicating a better family-provider alliance.
Ages & Stages: Social Emotional-2 | Baseline
  This Screener will evaluate 1-72 months old children in 7 areas of social-emotional development: self-regulation, compliance, social communication adaptive functioning, autonomy, affect, and interaction with people. Caregivers of children who score above threshold in the ASQ-SE will be eligible to participate in the study.
  Score range: 0-155 (the higher, the more concerning and to refer)
Emotion Dysregulation Inventory-Young Child | Baseline, immediately after intervention, and 3-months after intervention
  This is a 22-item tool for children aged 3-6 years to measure mental health symptoms of reactivity and dysphoria. 57point scale from "not at all" to "very severe".
  Higher scores generally indicate greater difficulties with emotion regulation.
Clinical Global Impression-Severity Scale | Baseline, immediately after intervention, and 3-months after intervention
  This is a 7-point scale to rate the severity of mental health symptoms.
  1: Normal, not at all ill. 2: Borderline mentally ill. 3: Mildly ill. 4: Moderately ill. 5: Markedly ill. 6: Severely ill. 7: Among the most extremely ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Kamimura-Nishimura, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No